CLINICAL TRIAL: NCT04607291
Title: Increasing Access and Developing Predictors for Colorectal Cancer Screening for Minority and Medicaid Clients
Brief Title: Health Service Intervention for the Improvement of Access and Adherence to Colorectal Cancer Screening
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: I 63518; NCI-2019-06075 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 63518 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH); R41CA232824 (NIH)
Record Dates: First submitted 2020-09-16; First posted 2020-10-29 (Actual); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Community Health Services

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health services research (Witness CARES services) Intervention (Experimental): Patients who are not prepared for a colonoscopy or stool test receive educational materials, messages, and videos electronically or by mail with information about colorectal screening and are followed up by phone within 2 weeks. Patients desiring colonoscopy, receive navigators assistance with obtaining the screening (e.g.,determining gastrointestinal doctor, scheduling appointment, prep materials and process, transportation, escort). Patients desiring a stool test, receive navigators assistance by facilitating fecal tests.
  Interventions: Other: Community Health Service; Other: Survey Administration

INTERVENTIONS:
Other: Community Health Service — Receive Witness CARES services
Other: Survey Administration — Ancillary studies

SUMMARY:
This phase I study investigates how well a health service program called Witness CARES Services works in increasing access and adherence to colorectal cancer screening in patients who have not undergone a colorectal screening in the past year. Providing patients with navigational and screening services via Witness CARES Services may improve access to and adherence levels of colorectal screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility of Witness CARES (WC) Services to achieve colorectal carcinoma (CRC) screening for non-adherent Medicaid clients.

II. Develop an algorithm for predicting CRC screening outcomes following intervention services.

OUTLINE:

Patients who are not prepared for a colonoscopy or stool test receive educational materials, messages, and videos electronically or by mail with information about colorectal screening and are followed up by phone within 2 weeks. Patients desiring colonoscopy receive navigator assistance with obtaining the screening (e.g.,determining gastrointestinal doctor, scheduling appointment, prep materials and process, transportation, escort). Patients desiring a stool test receive navigator assistance by facilitating fecal tests.

After completion of study, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are non-adherent to CRC screening over the past year (i.e., no stool testing in past 11 months or colonoscopy for over 9 years)
* Medicaid or Medicaid/Medicare subscribers
* Uninsured patients may be included from Mercy Comprehensive Care Center (MCCC), but will only be eligible for services to obtain fecal immunochemical tests (FIT) through the New York State (NYS) Cancer Services Program

Exclusion Criteria:

* Any participants from the lists of gaps in care clients from insurance or primary care practices who report having had a colonoscopy in the past 9 years (or having positive findings such as polyps, 5 years) or having completed some type of fecal test for CRC will be excluded
* Participants under 50 will be excluded unless they have been deemed high risk by their physician, and have a prescription for CRC screening
* Participants symptomatic for CRC will be excluded from the study

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2021-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Erwin, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Health Services Research (Witness CARES Services) Intervention
Started | 183
Completed | 183
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Health Services Research (Witness CARES Services) Intervention
Number analyzed (Participants) | 183
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 65
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 71
  White | 87
  More than one race | 0
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  United States | 183
Insurance Status [Count of Participants; unit: Participants]
  Medicare/Medicaid | 183
  non Medicare/Medicaid | 0
  Uninsured | 0
Screening Eligibility [Count of Participants; unit: Participants] — Does the participant meet the requirements/guidelines for CRC screening?
  Participants
    Eligible | 183
    non-Eligible | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Screening Metrics
Description: After CRC screening, satisfaction surveys will be conducted in order to assess the services of the Witness Cares Program.
  Below are responses to basic follow-up questions.
Time Frame: Up to 12 months
Population: There were a total of n=56 patients that received screening, of those patients, n=50 completed satisfaction surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Witness CARES Services) Intervention
Number analyzed (Participants) | 50
Participants
  Definitely helped me complete my CRC screening: Yes | 42
  Definitely helped me complete my CRC screening: No | 8
  Needed Education or Help with At Home Test: Yes | 37
  Needed Education or Help with At Home Test: No | 13
  Needed Reminder Calls: Yes | 33
  Needed Reminder Calls: No | 17
  Needed Help understanding CRC Screening Tests: Yes | 31
  Needed Help understanding CRC Screening Tests: No | 19
  Likely to Refer a Friend to Witness Cares Services: Yes | 45
  Likely to Refer a Friend to Witness Cares Services: No | 5

2. Primary Outcome: Model Development for Prediction of Intent and Colorectal Cancer (CRC) Screening Behaviors
Description: A telephone assessment of 118 self reported questions will be conducted in order to assess what factors are associated with CRC screening.
  The outcome of interest is CRC screening (colonoscopy or fecal immunochemical testing (FIT) test), which is treated as a binary outcome.
  The potential predictors include basic demographic characteristics as well as the survey sub-scales (based on the 118 self-reported questions).
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Witness CARES Services) Intervention
Number analyzed (Participants) | 183
Participants
  Screened | 56
  Not Screened | 127
Statistical Analysis 1: Comparison: Health Services Research (Witness CARES Services) Intervention; Test type: Other — A logistic regression model was used to identify factors associated with screening; A logistic regression model was used to identify factors associated with screening. A stepwise selection procedure (alpha entry and alpha exit = 0.15) was used to determine what factors were included in the model. Overall performance is assessed using the AUC. Factors included in the model: sex, stool test recommended by physician, know where to get stool test, fear of colonoscopy index score, ABR - afraid score, and knowledge that colonoscopy can reduce worry. AUC: 0.71

3. Secondary Outcome: Prediction of Which CRC Screening Test is Most Acceptable
Description: Data collected from surveys from the intent to screen clients will be used to help predict CRC screening test most acceptable
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Health Services Research (Witness CARES Services) Intervention
Number analyzed (Participants) | 183
Participants
  High Intent to Get Fit Test | 112
  Low Intent to get Fit Test | 71
  Unknown | 2
Statistical Analysis 1: Comparison: Health Services Research (Witness CARES Services) Intervention; Evaluating factors associated with high intent of getting a Fit test; Test type: Other — A logistic regression model was used to identify characteristics associated with high intent of getting a Fit test; A logistic regression model was used to identify factors associated with high intent of getting a fit test. A stepwise selection procedure (alpha entry and alpha exit = 0.15) was used to determine what factors were included in the model. Overall performance is assessed using the AUC. Factors included in the model: sex, race, stool test or colonoscopy recommended by physician, know where to get stool test, CBPR score, and barriers to screening score. AUC: 0.80

ADVERSE EVENTS:
Time Frame: 30 days post contact with navigator.
Arm/Group | Health Services Research (Witness CARES Services) Intervention
All-Cause Mortality (participants affected / at risk) | 0/183
Serious Adverse Events (participants affected / at risk) | 0/183
Other Adverse Events (participants affected / at risk) | 0/183

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04607291/Prot_SAP_000.pdf